CLINICAL TRIAL: NCT04535362
Title: Impact of Menthol on the Abuse Potential of Nicotine
Brief Title: Nicotine's Potential Abuse With Menthol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000029223; 2U54DA036151-06 (NIH)
Record Dates: First submitted 2020-08-24; First posted 2020-09-01 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: subjects will be unblinded to smoking menthol or non menthol for two weeks before each test session. Each session will include 3 infusions in the same order: nicotine (1 mg per 70 kg body weight) delivered over 5 minutes, saline and nicotine (1 mg/ 70 kg) delivered over 2.5 minutes. Once the participants complete the test session, participants will be crossed-over to the alternative treatment.
Who Masked: Participant
Masking Description: The cigarette condition is unblinded but the nicotine infusion is blinded to participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- menthol cigarettes (Active Comparator): Will smoke only menthol cigarettes for two weeks
  Interventions: Drug: Nicotine
- non menthol cigarettess (Active Comparator): Will only smoke non menthol cigarettes for two weeks
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — session will include 3 infusions in the same order: nicotine (1 mg per 70 kg body weight) delivered over 5 minutes, saline and nicotine (1 mg/ 70 kg) delivered over 2.5 minutes.
  Other Names: intravenous nicotine

SUMMARY:
To examine if switching from menthol to non-menthol cigarettes will change the dose-effect curves for positive subjective effects and alleviation of smoking urges as a function of nicotine delivery rate in smokers.

DETAILED DESCRIPTION:
A placebo-controlled study that will recruit male and female menthol nicotine dependent smokers. Following screening and evaluation as described above, eligible participants will be enrolled in the study which will last about 4 weeks. Eligible, participants will be randomized to menthol or non-menthol smoking condition for 2 weeks (Phase 1) and then will be switched to the alternative condition for another 2 weeks (Phase 2). The smoking condition will be open label. Participants will be provided with free cigarettes in Phases 1 and 2. For the menthol condition, participants will be provided their usual brand of menthol cigarettes and for the non-menthol condition, they will be provided a matched-brand non-menthol cigarette (e.g., Newport Non-Menthol Gold 100s for those who smoke Newport Menthol Gold 100s). In week 2 of each Phase, participants will have a test session. Each session will include 3 infusions in the same order: nicotine (1 mg per 70 kg body weight) delivered over 5 minutes, saline and nicotine (1 mg/ 70 kg) delivered over 2.5 minutes. Once the participants complete the test session, participants will be crossed-over to the alternative treatment. The period between the 2 Phases will not be longer than one week.

ELIGIBILITY:
Inclusion Criteria:

* 1) Female and male smokers, aged 21 to 35 years, who have been smoking tobacco cigarettes for at least a year;
* 2) smoke ≥ 5 and less than 20 cigarettes per day;
* 3) urine cotinine levels > 100 ng/mL consistent with nicotine intake of an active smoker
* 4) not seeking treatment at the time of the study for nicotine dependence;
* 5) in good health as verified by medical history, screening examination, and screening laboratory tests;
* 6) for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* 1) history of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the subject to be in the study;
* 2) regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics);
* 3) current alcohol or substance dependence for any other recreational or prescription drugs other than nicotine;
* 4) use of e-cigarettes more than 10 days in the past 30 days;
* 5) urine drug screening indicating recent illicit drugs use (with the exception of marijuana).

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs Hospital, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Menthol FIRST, Non-Menthol SECOND; Non-Menthol FIRST, Menthol SECOND: Participants were randomized to either menthol or non-menthol cigarette smoking condition for 2 weeks (Phase 1) and then switched to the other condition for another 2 weeks (Phase 2), in a crossover design. Participants received free cigarettes throughout both phases.
Period: Overall Study
Arm/Group | Menthol FIRST, Non-Menthol SECOND | Non-Menthol FIRST, Menthol SECOND
Started | 8 | 8
Entered Phase 1 | 8 | 8
Completed Phase 1 | 8 | 8
Entered Phase 2 | 8 | 8
Completed Phase 2 | 5 | 7
Completed | 5 | 7
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: Participants randomized to one of two crossover arms.
Groups:
- Study Participants: All participants in the study prior to randomization to crossover order. Eligible participants were individuals who reported smoking at least 5 cigarettes a day for the past year and had urine cotinine levels exceeding 100 ng/mL, an indicator of daily smoking. Participants were not interested in quitting smoking and were free of major medical and psychiatric disorders, including substance use disorders (except tobacco use), as confirmed by medical and psychiatric assessment.
Arm/Group | Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Average number of cigarettes consumed daily [Mean (Standard Deviation); unit: cigarettes per day] | 10.5 (4.7)
Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: units on a scale] — The total score ranges from 0 to 10. Higher scores indicate a greater dependence on nicotine:
  0-2 points: Very low dependence, 3-4 points: Low dependence, 5 points: Medium dependence, 6-7 points: High dependence, 8-10 points: Very high dependence.
  units on a scale | 4.2 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Drug Effect Questionnaire - Stimulatory Effects
Description: Drug Effects Questionnaire was used to assess participants. The DEQ is consist of 10 items measured on a 1 to 100 visual analog scale, ranging from "not at all" to "extremely.". These ratings were then averaged to create three domain scores reflecting 1) stimulatory effects (average of "feel stimulated", "feel drug effects" and "feel high"), 2) pleasurable effects (average of "like", "feel good " and "want more"), and 3) aversive effects (average of "feel anxious", "feel down" and "feel bad"). Head rush was also assessed. Scores on the subscales range from 0 - 100 where 0 is the measure of least impactful 'effect'.
Time Frame: Following 2 weeks of smoking, the procedure took over 3 hours, with measured effects at 2.5 minutes, 5 minutes and 10 minutes
Population: Participants assessed an any or both points in the crossover design.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Menthol; Non-Menthol: Participants were randomized to either menthol or non-menthol cigarette smoking condition for 2 weeks (Phase 1) and then switched to the other condition for another 2 weeks (Phase 2), in a crossover design. Participants received free cigarettes throughout both phases.
Arm/Group | Menthol | Non-Menthol
Number analyzed (Participants) | 16 | 13
units on a scale
  2.5 Minutes | 39.37 (24.41) | 33.48 (19.73)
  5 minutes | 32.35 (27.93) | 33.23 (28.79)
  10 minutes | 13.19 (16.15) | 19.43 (21.41)
Statistical Analysis 1: Comparison: Menthol vs Non-Menthol; The fixed effects in the mixed models were infusion rate (2.5 minutes, 5 minutes and 10 minutes (placebo)), cigarette condition (menthol vs. non-menthol), and their interaction. We also controlled for order effects of cigarette condition by including session in the models Subject was a clustering factor and different variance-covariance structures were considered within each condition and subject. The best-fitting structure was selected based on Schwartz's Bayesian Criterion; Test type: Superiority; p = 0.93, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.63

2. Primary Outcome: Drug Effect Questionnaire - Pleasure Effect
Description: Drug Effects Questionnaire was used to assess participants. The DEQ is consist of 10 items measured on a 1 to 100 visual analog scale, ranging from "not at all" to "extremely.". These ratings were then averaged to create three domain scores reflecting: 1) stimulatory effects (average of "feel stimulated", "feel drug effects" and "feel high"), 2) pleasurable effects (average of "like", "feel good " and "want more"), and 3) aversive effects (average of "feel anxious", "feel down" and "feel bad"). Head rush was also assessed. Scores on the subscales range from 0 - 100 where 0 is the measure of least impactful 'effect'.
Time Frame: as for outcome 1
Population: Participants assessed an any or both points in the crossover design.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol | Non-Menthol
Number analyzed (Participants) | 16 | 13
units on a scale
  2.5 minutes | 37.51 (28.35) | 27.25 (17.62)
  5 minutes | 36.49 (31.55) | 29.28 (25.42)
  10 minutes | 23.42 (20.80) | 24.71 (18.37)
Statistical Analysis 1: Comparison: Menthol vs Non-Menthol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.68, Mixed Models Analysis; Mean Difference (Net) = 0.12, Standard Error of Mean 0.30

3. Secondary Outcome: SAFTEE
Description: The SAFTEE is a technique for the systematic assessment of side effects in clinical trials developed by National Institute of Mental Health. It is a questionnaire that rates the current severity of a wide range of somatic, behavioral and affective symptoms in general and specific inquiry formats. It is designed to report adverse health events, regardless of whether or not they are suspected to be drug related, in order to reduce the under-reporting of unanticipated events compared with "known or expected" events.
Time Frame: up to one year
Population: these data were not collected
Arm/Group | Menthol Cigarettes | Non Menthol Cigarettess
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Drug Effect Questionnaire - Aversive Effect
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Participants assessed an any or both points in the crossover design.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol | Non-Menthol
Number analyzed (Participants) | 16 | 13
units on a scale
  2.5 minutes | 11.33 (11.78) | 14.76 (15.56)
  5 minutes | 8.73 (11.12) | 11.23 (13.78)
  10 minutes | 6.33 (8.50) | 6.92 (8.79)
Statistical Analysis 1: Comparison: Menthol vs Non-Menthol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Net) = 0.46, Standard Error of Mean 0.51

5. Primary Outcome: Drug Effect Questionnaire - Head Rush
Description: Drug Effects Questionnaire was used to assess participants. The DEQ is consist of 10 items measured on a 1 to 100 visual analog scale, ranging from "not at all" to "extremely.". These ratings were then averaged to create three domain scores reflecting: 1) stimulatory effects (average of "feel stimulated", "feel drug effects" and "feel high"), 2) pleasurable effects (average of "like", "feel good " and "want more"), and 3) aversive effects (average of "feel anxious", "feel down" and "feel bad"). Head rush was also assessed. Scores on all subscales, including Head Rush scale, range from 0 - 100 where lower scores indicate less head rush.
Time Frame: as for outcome 1
Population: Participants assessed an any or both points in the crossover design.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol | Non-Menthol
Number analyzed (Participants) | 16 | 13
units on a scale
  2.5 minutes | 31.73 (32.55) | 14.76 (15.56)
  5 minutes | 19.20 (25.48) | 11.23 (13.78)
  10 minutes | 8.93 (13.93) | 6.92 (8.79)
Statistical Analysis 1: Comparison: Menthol vs Non-Menthol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Net) = 1.26, Standard Error of Mean 0.98

ADVERSE EVENTS:
Time Frame: 4 weeks total (2 sessions of 2 week smoking periods) - each with 2 3 hour sessions.
Arm/Group | Menthol | Non-Menthol
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/16 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04535362/Prot_SAP_000.pdf